CLINICAL TRIAL: NCT04981210
Title: National Taiwan University Hospital
Brief Title: High Risk Screen of Childhood Late-onset Pompe Disease in Pediatric Outpatient Clinics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012243RIPC
Record Dates: First submitted 2021-07-07; First posted 2021-07-28 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-08

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspect LOPD

SUMMARY:
Establish of high-risk screening criteria to earlier identify possible childhood LOPD for early treatment and better prognosis. Therefore, validation of the high-risk screening criteria for childhood LOPD will be critical for identifying children of LOPD in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Children who are >1 year and < 18 year of age from pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH

Exclusion Criteria:

* Children who have been diagnosed as specific neuromuscular disorders.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects who are >1 year and < 18 year of age will be enrolled from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
clinical signs/symptoms surveyed - Weakness in neck (No.1) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
clinical signs/symptoms surveyed - Symptoms and signs of muscle weakness (No.2) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
  Symptoms and signs of muscle weakness including Frequent fall, difficulty to climb stairs, poor performance in physical education classes, gait abnormalities or facial weakness.
clinical signs/symptoms surveyed - Unable to speak clearly / keep slobbering (No.3) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
clinical signs/symptoms surveyed - Scoliosis (No.4) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
clinical signs/symptoms surveyed - Motor developmental delay (No.5) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
clinical signs/symptoms surveyed - Persist diarrhea with unknown cause (No.6) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
clinical signs/symptoms surveyed - Frequent respiratory infections (No.7) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
clinical signs/symptoms surveyed - Morning headache (No.8) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
clinical signs/symptoms surveyed - Urinary / Fecal incontinence (No.9) | 2 years
  Children from outpatient clinics of pediatric neurology, pediatric orthopedics and pediatric rehabilitation in NTUH will be surveyed whether they have clinical signs/symptoms. Any patients who fulfill symptom No. 1 or 3 associated to the difficulty of flexing the neck from supine position or accumulated 3 findings from pediatric orthopedics and pediatric rehabilitation will be referred to pediatric neurology for double confirmation that patients meet the criteria.
dry blood sample (DBS) - GAA activity analysis | 2 years
  Then we will use dry blood sample (DBS) or whole blood sample for screening the possibility of Pompe disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-Chin Weng, Taipei, Taiwan